CLINICAL TRIAL: NCT01506960
Title: Evaluation of a Combined Near Infrared Spectroscopy (NIRS) and Intravascular Ultrasound (IVUS) Catheter for Detection of Lipid Rich Plaque
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: It was felt that a sufficient number of subjects were enrolled.
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Infraredx (Industry)
Responsible Party: Principal Investigator, Ik-Kyung Jang, MD, PhD, Professor of Medicine, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2010P001608
Record Dates: First submitted 2012-01-03; First posted 2012-01-10 (Estimated); Results first posted 2013-10-18 (Estimated); Last update posted 2013-11-18 (Estimated); Status verified 2013-10

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Coronary stenting with OCT, NIRS/IVUS (Experimental): All subjects will have Near Infrared Spectroscopy/Intravascular Ultrasound Imaging performed.
  Interventions: Device: InfraReDx Lipiscan IVUS

INTERVENTIONS:
Device: InfraReDx Lipiscan IVUS — Near Infrared Spectroscopy/Intravascular Ultrasound will be performed following OCT imaging.

SUMMARY:
The purpose of this study is to learn more about lipid rich plaque using Near Infrared Spectroscopy (NIRS)/Intravascular Ultrasound (IVUS) imaging in patients who have had coronary artery stenting and Optical coherence tomography (OCT) imaging.

DETAILED DESCRIPTION:
The aims of this study are to:

1. Test the ability of the new NIRS IVUS system to detect lipid pool
2. Evaluate the accuracy of the NIRS IVUS system for localization of lipide rich plaque: superficial vs deep
3. Improve diagnostic accuracy of OCT for detection of lipid using information from NIRS IVUS

ELIGIBILITY:
Inclusion Criteria:

Patient Characteristics

1. Males and non-pregnant females > 18 and < 79 years of age
2. Patients referred for diagnostic coronary angiography who are found to have lesions in native coronary arteries which will be treated by percutaneous coronary intervention (PCI) (or patients with known coronary lesions who are referred for planned PCI)
3. Able to give written informed consent

Lesion Characteristics

1. Lesion in native coronary artery
2. Angiographic stenosis > 50%
3. Reference vessel diameter 2.5 mm - 4.0 mm by visual estimation
4. Subjects who have successful PCI and OCT

General Exclusion Criteria

1. Subjects who are unable or unwilling to sign the informed consent form
2. Subjects with serious co-morbid conditions that in judgment of the investigator preclude inclusion in this study (such as terminal cancer, life expectancy < 6 months, Liver Function Tests (LFTs) > 3 times Upper Limit of Normal (ULN), or post-transplant)
3. Subjects with New York Heart Association (NYHA) class III or IV heart failure or known left ventricular ejection fraction < 30%
4. Subjects who have experienced an ST-elevation myocardial infarction (STEMI) within 72 hours prior to the procedure
5. Subjects with hemodynamic or electrical instability (including shock)
6. Subjects diagnosed with severe, non-catheter-related coronary artery spasm
7. Subjects who are or may be pregnant
8. Subjects with known allergies to contrast media
9. Subjects with renal failure as defined by estimated Glomerular Filtration Rate (eGFR) < 60.
10. History of Transient Ischemic Attack (TIA) or stroke < 6 months

Lesion Specific Exclusion Criteria These exclusion criteria apply to the target lesion to be imaged by NIRS IVUS.

1. Lesion located in the left main coronary artery
2. Lesions that are heavily calcified
3. Lesions where OCT cannot be performed due to technical difficulties
4. Other lesions that the investigator deems inappropriate for the procedure such as lesions with excessive tortuosity, presence of thrombus, low flow by TIMI grade.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2012-01; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ik-Kyung Jang, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Coronary Stenting With OCT, NIRS/IVUS
Started | 64
Completed | 17
Not Completed | 47
Not completed — Did not meet angiographic criteria | 47

BASELINE CHARACTERISTICS:
Population: 47 subjects did not meet angiographic criteria for participation.
Arm/Group | Subjects Having NIRS/IVUS and OCT Imaging During PCI.
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 5
Age Continuous [Mean (Standard Deviation); unit: years] | 59.8 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 14
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Detection of Lipid Rich Plaque by Near Infrared Spectroscopy (NIRS) Intravascular Ultrasound (IVUS)
Description: Subjects are presenting for their clinically-indicated cardiac catheterization. NIRS/IVUS imaging will be done at the time of catheterization.
Time Frame: Measured one point in time during cardiac catheterization
Measure: Number; unit: % pts with lipid on NIRS and OCT
Arm/Group | Subjects Having NIRS/IVUS and OCT Imaging During PCI.
Number analyzed (Participants) | 17
% pts with lipid on NIRS and OCT | 90

2. Secondary Outcome: Differences in NIRS Parameters Between Deep and Superficial Lipid Assessed by Optical Coherence Tomography (OCT).
Description: Subjects are presenting for their clinically-indicated cardiac catheterization. NIRS/IVUS imaging will be done at the time of catheterization. Plaques were divided depending on depth of lipid by OCT (cut off value 130 um).
Time Frame: Measured at the time of cardiac catheterization
Population: Per protocol
Measure: Mean (Standard Deviation); unit: mm (LCP length)
Units Other Than Participants: Lesions
Arm/Group | Superficial Lipid | Deep Lipid
Number analyzed (Participants) | 6 | 5
Number analyzed (Lesions) | 9 | 9
mm (LCP length) | 5.5 (2.8) | 4.1 (3.1)

ADVERSE EVENTS:
Arm/Group | Subjects Having NIRS/IVUS and OCT Imaging During PCI.
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 5/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects Having NIRS/IVUS and OCT Imaging During PCI. (N=17)
Back pain post procedure (Musculoskeletal and connective tissue disorders) | 2 (2)
Non-ischemic chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Post-procedural myocardial infarction (Cardiac disorders) | 1 (1)
PVCs during NIRS IVUS (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes